CLINICAL TRIAL: NCT01270087
Title: The Effect of Adalimumab (Humira) on Vascular Abnormalities in Rheumatoid Arthritis. A Pilot Study.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Abbott (Industry); The Swedish Research Council (Other Government); The Swedish Rheumatism Ass (Other); Crafoord Foundation (Other)
Responsible Party: Carl Turesson, Associate Professor, Department of Rheumatology, Skåne University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REUMAUMAS 2005-1; 2005-000129-47 (EudraCT Number)
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis, cardiovascular disease, adalimumab
MeSH Terms: conditions — Arthritis, Rheumatoid; Cardiovascular Diseases | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adalimumab (Other)
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — 40 mg IV every 14 days
  Other Names: Humira

SUMMARY:
The purpose of this study is to determine whether anti-inflammatory treatment with adalimumab (Humira) reduces endothelial activation in blood vessels in patients with active rheumatoid arthritis. Markers of endothelial activation are assessed in muscle tissue before treatment and after 3 months, and related to other biomarkers and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rheumatoid arthritis
* Fulfillment of the American College of Rheumatology 1987 criteria for rheumatoid arthritis
* Active disease despite treatment with at least one disease modifying anti-rheumatic drug
* Treatment with adalimumab indicated according to the the patient's rheumatologist
* At least six swollen joints in 28-joint index
* CRP > 8 mg / L within the last three months

Exclusion Criteria:

* Treatment with anti-TNF drugs in the last three months
* Treatment with intravenous corticosteroids within fourteen days
* Ongoing treatment with oral high-dose corticosteroids (equivalent to ≥ 20 mg of prednisolon daily) or completed such treatment less than fifteen days before inclusion
* Severe bleeding disorder
* Extensive or refractory leg ulcers
* Severe peripheral vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Endothelial expression of HLA-DQ in muscle biopsies | 3 months
  Vascular tissue area stained for HLA-DQ by immunohistochemistry, quantified by computer assisted image analysis
Endothelial expression of interleukin-1 alpha in muscle biopsies | 3 months
  Vascular tissue area stained for interleukin-1 alpha by immunohistochemistry, quantified by computer assisted image analysis
Carotid artery intima-media thickness | 3 months
  Thickness of the intima and media of the common carotid artery, measured by ultrasound. Mean of two measures of the right and left common carotid artery.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Turesson, MD, PhD, Principal Investigator — Department of Rheumatology, Skåne University Hospital
Locations (1):
- Department of Rheumatology, Skåne University Hospital, Malmo, Sweden